CLINICAL TRIAL: NCT05291780
Title: STereotactic Ablative RadioTherapy in NEWly Diagnosed and Recurrent Locally Advanced Non-small Cell Lung Canter Patients Unfit for concurrEnt RAdio-chemotherapy
Brief Title: Stereotactic Ablative Radiotherapy in Locally Advanced Non Small Cell Lung Cancer
Acronym: START-NEW-ERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radiotherapy Oncology Centre "Santa Maria" Hospital (Other)
Collaborators: Paola Anselmo,MD (Unknown); Michelina Casale,PhD (Unknown); Ernesto Maranzano,MD (Unknown); Fabio Trippa,MD (Unknown)
Responsible Party: Principal Investigator, Fabio Arcidiacono, MD, Principal Investigator, Radiotherapy Oncology Centre "Santa Maria" Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SABR-LA-NSCLC 810
Record Dates: First submitted 2022-03-07; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma
Keywords: LA-NSCLC; SABR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SABR in unresectable LA-NSCLC (Experimental): Patients fit for chemotherapy will be enrolled to sequential chemotherapy-stereotactic ablative radiotherapy (SABR), while patients unfit for chemotherapy will be enrolled to exclusive stereotactic ablative radiotherapy (SABR).
  Interventions: Radiation: Stereotactic Ablative Radiotherapy in Unresectable Locally Advanced Non-Small Cell Lung Cancer

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy in Unresectable Locally Advanced Non-Small Cell Lung Cancer — The prescribed dose of stereotactic ablative radiotherapy (SABR) will be of at least 35-40 Gy in 5 fractions. The dose of SABR will be increased, case by case, respecting the maximum tolerance dose of the healthy structures.
  Participants will SABR once a day for 5 days, Monday through Friday (around 1 week).

SUMMARY:
This is a prospective, non-randomized, single arm, single institution phase II trial to evaluate the safety and effectiveness of stereoractic ablative radiotherapy (SABR) in selected unresectable newly diagnosed and recurrent locally advanced (LA) non-small cell lung cancer (NSCLC) patients unfit for concurrent chemo-radiotherapy (ChT-RT).

Patients unfit for concurrent ChT-RT but fit for chemotherapy will be enrolled to sequential ChT-SABR; patients unfit for ChT will be enrolled to exclusive SABR.

DETAILED DESCRIPTION:
Current standard of care for fit patients with unresectable LA-NSCLC is concurrent chemo-radiotherapy (ChT-RT) which consists of 6 weeks of radiation and chemotherapy. Unfortunately many LA NSCLC patients, particularly the elderly, are unfit for concurrent ChT-RT because of their poor performance status and co-morbidities. Sequential ChT-RT and/or exclusive RT are options available for patients not suitable for concomitant approaches.

Median progression-free survival among patients receiving concurrent ChT-RT is poor and no more than 15% of cases are alive at 5 years.

This study is evaluating SABR in unresectable LA-NSCLC. Hypofractionated regimens of RT have emerged as a possible approach in LA-NSCLC, not only because prolonged treatments may discourage a proportion of elderly patients (20-30%) who are forced to give up treatment due to distance from the Radiotherapy Centre, but also for radiobiological reasons.

Recent technological advances in RT, first of all stereotactic body radiotherapy (SBRT), have made hypofractionation widely applicable with the possibility to administer few (5 to 8) fractions of high external beam doses to the tumor, sparing the surrounding healthy tissues by a rapid fall of dose outside the target.

LA-NSCLC patients will be discussed at the multidisciplinary lung cancer group and will be judged unfit for surgery and concurrent ChT-RT (e.g. elderly patients and/or large volume of disease and/or cardiovascular comorbidities) but suitable for RT. Neoadjuvant ChT will be evaluated case by case and will be prescribed only in fit patients.

Starting from the standard radical conventionally administered dose for LA-NSCLC (equivalent to at least 54-60 Gy in 27-30 fractions), the investigators decided to prescribe an ablative dose of at least 35-40 Gy in 5 fractions.

The SABR dose will be increased, case by case, respecting the maximum tolerance dose of healthy structures.

The purpose of this study is to explore SABR in the treatment of unresectable LA-NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Histologically or cytologically confirmed non-small cell lung cancer
* LA-NSCLC at the first diagnosis or recurrent LA-NSCLC after previous surgery
* Stage II-III disease as determined by PET/CT and TC/MRI Brain (American Joint Committee on Cancer 7th or 8th Edition)
* oligo-metastatic LA-NSCLC with metastasis suitable to local treatment in the primary and metastatic site
* Participant is not eligible for surgical resection as determined by the multidisciplinary lung cancer group
* Participant is not eligible for concurrent chemotherapy as determined by the multidisciplinary lung cancer group
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* LA-NSCLC patients eligible for surgical resection
* ECOG performance status 3 or more
* Inability to safely treat target lesions
* Pregnant women are excluded from this study because radiation therapy has known potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Local control | 1 year, 2 years and 3 years
  A lack of progression (i.e., any response and stable disease) of the treated volume according to RECIST and PERCIST. Local recurrence (LR) was defined as tumor progression within the radiation field (95% of the recurrence volume within the original 80% isodose of SABR). Local recurrence-free survival (LR-FS) was defined as the interval between treatment and radiological evidence of LR.
Proportion of Participants Experiencing Grade 3 or Higher Toxicities | 6 months and 1 year
  SABR will be considered safe if no grade (G) 3 or higher toxicities appears. Toxicity, graded according to Common Terminology Criteria for Adverse Events (CTCAE v3.0) will be assessed during SABR and at all follow-up intervals. Toxicity will be recorded as acute when occurred during SABR or within 3 months after completion of treatment. When the time interval will be longer than 3 months, toxicity will be defined late.

SECONDARY OUTCOMES:
Thoracic nodal-recurrence free survival | 1 year, 2 years and 3 years
  The interval between treatment and radiological evidence of any nodal recurrence outside the treated nodes and anyway outside the original isodose of 80%
Distant progression free-survival | 1 year, 2 years and 3 years
  The interval between treatment and radiological evidence of systemic disease progression
Overall Survival | 1 year, 2 years, 3 years and 5 years
  The overall survival will be calculated from treatment to patient death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Arcidiacono, MD, Principal Investigator — Radiotherapy Oncology Centre "S.Maria" Hospital; Paola Anselmo, MD, Principal Investigator — Radiotherapy Oncology Centre "S.Maria" Hospital; Michelina Casale, PhD, Principal Investigator — Radiotherapy Oncology Centre "S.Maria" Hospital; Fabio Trippa, MD, Study Director — Radiotherapy Oncology Centre "S.Maria" Hospital; Ernesto Maranzano, MD, Study Chair — Radiotherapy Oncology Centre "S.Maria" Hospital
Locations (1):
- Radiotherapy Oncology Centre "S.Maria" Hospital, Terni, TR, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang S, Wong ML, Hamilton N, Davoren JB, Jahan TM, Walter LC. Impact of age and comorbidity on non-small-cell lung cancer treatment in older veterans. J Clin Oncol. 2012 May 1;30(13):1447-55. doi: 10.1200/JCO.2011.39.5269. Epub 2012 Mar 26. PMID 22454424
- [Result] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Result] De Ruysscher D, Botterweck A, Dirx M, Pijls-Johannesma M, Wanders R, Hochstenbag M, Dingemans AM, Bootsma G, Geraedts W, Simons J, Pitz C, Lambin P. Eligibility for concurrent chemotherapy and radiotherapy of locally advanced lung cancer patients: a prospective, population-based study. Ann Oncol. 2009 Jan;20(1):98-102. doi: 10.1093/annonc/mdn559. Epub 2008 Aug 20. PMID 18718891
- [Result] Sigel K, Lurslurchachai L, Bonomi M, Mhango G, Bergamo C, Kale M, Halm E, Wisnivesky J. Effectiveness of radiation therapy alone for elderly patients with unresected stage III non-small cell lung cancer. Lung Cancer. 2013 Nov;82(2):266-70. doi: 10.1016/j.lungcan.2013.06.011. Epub 2013 Sep 5. PMID 24011407
- [Result] Rodrigues G, Choy H, Bradley J, Rosenzweig KE, Bogart J, Curran WJ Jr, Gore E, Langer C, Louie AV, Lutz S, Machtay M, Puri V, Werner-Wasik M, Videtic GMM. Definitive radiation therapy in locally advanced non-small cell lung cancer: Executive summary of an American Society for Radiation Oncology (ASTRO) evidence-based clinical practice guideline. Pract Radiat Oncol. 2015 May-Jun;5(3):141-148. doi: 10.1016/j.prro.2015.02.012. PMID 25957184
- [Result] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Result] Fowler JF, Chappell R. Non-small cell lung tumors repopulate rapidly during radiation therapy. Int J Radiat Oncol Biol Phys. 2000 Jan 15;46(2):516-7. doi: 10.1016/s0360-3016(99)00364-8. No abstract available. PMID 10661362
- [Result] Belderbos J, Walraven I, van Diessen J, Verheij M, de Ruysscher D. Radiotherapy dose and fractionation for stage III NSCLC. Lancet Oncol. 2015 Apr;16(4):e156-7. doi: 10.1016/S1470-2045(15)70121-X. No abstract available. PMID 25846093
- [Result] David EA, Daly ME, Li CS, Chiu CL, Cooke DT, Brown LM, Melnikow J, Kelly K, Canter RJ. Increasing Rates of No Treatment in Advanced-Stage Non-Small Cell Lung Cancer Patients: A Propensity-Matched Analysis. J Thorac Oncol. 2017 Mar;12(3):437-445. doi: 10.1016/j.jtho.2016.11.2221. Epub 2017 Jan 18. PMID 28109804
- [Result] Kaster TS, Yaremko B, Palma DA, Rodrigues GB. Radical-intent hypofractionated radiotherapy for locally advanced non-small-cell lung cancer: a systematic review of the literature. Clin Lung Cancer. 2015 Mar;16(2):71-9. doi: 10.1016/j.cllc.2014.08.002. Epub 2014 Sep 28. PMID 25450876
- [Result] Kong C, Zhu X, Shi M, Wang L, Chen C, Tao H, Jiang N, Yan P, Zhao L, Song X, He X. Survival and Toxicity of Hypofractionated Intensity Modulated Radiation Therapy in 4 Gy Fractions for Unresectable Stage III Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):710-719. doi: 10.1016/j.ijrobp.2020.03.038. Epub 2020 Apr 7. PMID 32275994
- [Result] Franks KN, Jain P, Snee MP. Stereotactic ablative body radiotherapy for lung cancer. Clin Oncol (R Coll Radiol). 2015 May;27(5):280-9. doi: 10.1016/j.clon.2015.01.006. Epub 2015 Mar 4. PMID 25746732
- [Result] Arcidiacono F, Aristei C, Marchionni A, Italiani M, Fulcheri CPL, Saldi S, Casale M, Ingrosso G, Anselmo P, Maranzano E. Stereotactic body radiotherapy for adrenal oligometastasis in lung cancer patients. Br J Radiol. 2020 Nov 1;93(1115):20200645. doi: 10.1259/bjr.20200645. Epub 2020 Sep 2. PMID 32822540
- [Result] Bezjak A, Paulus R, Gaspar LE, Timmerman RD, Straube WL, Ryan WF, Garces YI, Pu AT, Singh AK, Videtic GM, McGarry RC, Iyengar P, Pantarotto JR, Urbanic JJ, Sun AY, Daly ME, Grills IS, Sperduto P, Normolle DP, Bradley JD, Choy H. Safety and Efficacy of a Five-Fraction Stereotactic Body Radiotherapy Schedule for Centrally Located Non-Small-Cell Lung Cancer: NRG Oncology/RTOG 0813 Trial. J Clin Oncol. 2019 May 20;37(15):1316-1325. doi: 10.1200/JCO.18.00622. Epub 2019 Apr 3. PMID 30943123
- [Result] Karam SD, Horne ZD, Hong RL, McRae D, Duhamel D, Nasr NM. Hypofractionated stereotactic body radiation therapy for elderly patients with stage IIB-IV nonsmall cell lung cancer who are ineligible for or refuse other treatment modalities. Lung Cancer (Auckl). 2014 Oct 3;5:59-66. doi: 10.2147/LCTT.S66395. eCollection 2014. PMID 28210143
- [Result] Schwartz LH, Litiere S, de Vries E, Ford R, Gwyther S, Mandrekar S, Shankar L, Bogaerts J, Chen A, Dancey J, Hayes W, Hodi FS, Hoekstra OS, Huang EP, Lin N, Liu Y, Therasse P, Wolchok JD, Seymour L. RECIST 1.1-Update and clarification: From the RECIST committee. Eur J Cancer. 2016 Jul;62:132-7. doi: 10.1016/j.ejca.2016.03.081. Epub 2016 May 14. PMID 27189322
- [Result] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Result] Nguyen NP, Bishop M, Borok TJ, Welsh J, Hamilton R, Cohen D, Nguyen LM, Vincent VH. Pattern of failure following chemoradiation for locally advanced non-small cell lung cancer: potential role for stereotactic body radiotherapy. Anticancer Res. 2010 Mar;30(3):953-61. PMID 20393019
- [Result] Faivre-Finn C, Vicente D, Kurata T, Planchard D, Paz-Ares L, Vansteenkiste JF, Spigel DR, Garassino MC, Reck M, Senan S, Naidoo J, Rimner A, Wu YL, Gray JE, Ozguroglu M, Lee KH, Cho BC, Kato T, de Wit M, Newton M, Wang L, Thiyagarajah P, Antonia SJ. Four-Year Survival With Durvalumab After Chemoradiotherapy in Stage III NSCLC-an Update From the PACIFIC Trial. J Thorac Oncol. 2021 May;16(5):860-867. doi: 10.1016/j.jtho.2020.12.015. Epub 2021 Jan 19. PMID 33476803
- [Result] Ahmed N, Hasan S, Schumacher L, Colonias A, Wegner RE. Stereotactic body radiotherapy for central lung tumors: Finding the balance between safety and efficacy in the "no fly" zone. Thorac Cancer. 2018 Oct;9(10):1211-1214. doi: 10.1111/1759-7714.12764. Epub 2018 Aug 10. PMID 30095228
- [Result] Nguyen KNB, Hause DJ, Novak J, Monjazeb AM, Daly ME. Tumor Control and Toxicity after SBRT for Ultracentral, Central, and Paramediastinal Lung Tumors. Pract Radiat Oncol. 2019 Mar;9(2):e196-e202. doi: 10.1016/j.prro.2018.11.005. Epub 2018 Nov 26. PMID 30496842
- [Result] Tekatli H, Haasbeek N, Dahele M, De Haan P, Verbakel W, Bongers E, Hashemi S, Nossent E, Spoelstra F, de Langen AJ, Slotman B, Senan S. Outcomes of Hypofractionated High-Dose Radiotherapy in Poor-Risk Patients with "Ultracentral" Non-Small Cell Lung Cancer. J Thorac Oncol. 2016 Jul;11(7):1081-9. doi: 10.1016/j.jtho.2016.03.008. Epub 2016 Mar 21. PMID 27013408
- [Derived] Arcidiacono F, Anselmo P, Casale M, Zannori C, Ragusa M, Mancioli F, Marchetti G, Loreti F, Italiani M, Bracarda S, Maranzano E, Trippa F. STereotactic Ablative RadioTherapy in NEWly Diagnosed and Recurrent Locally Advanced Non-Small Cell Lung Cancer Patients Unfit for ConcurrEnt RAdio-Chemotherapy: Early Analysis of the START-NEW-ERA Non-Randomised Phase II Trial. Int J Radiat Oncol Biol Phys. 2023 Mar 15;115(4):886-896. doi: 10.1016/j.ijrobp.2022.10.025. Epub 2022 Oct 24. PMID 36288758